CLINICAL TRIAL: NCT00977249
Title: Varenicline for Long-term Nicotine Replacement Therapy (NRT) Users. A Double Blind, Placebo Controlled Trial
Brief Title: Varenicline for Long-term Nicotine Replacement Therapy (NRT) Users
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Chief Physician Philip Tønnesen, M.D., Gentofte University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCTnumber 2008-006426-24
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Tobacco Dependence
Keywords: long term nicotine gum use; varenicline; adverse effects
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Palliative Care; Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Active Comparator): Varenicline for 12 weeks.
  The treatment schedule for varenicline is:
  Varenicline tablets, 0.5 mg x 1 daily, day 1-3 Varenicline 0.5 mg x 2, day 4-6 Varenicline 1 mg x 2, day 7 up to 12 weeks
  Interventions: Behavioral: support and visits; Drug: varenicline
- placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Behavioral: support and visits; Drug: placebo

INTERVENTIONS:
Behavioral: support and visits — visits at weeks 0,2,4,6,9 and 12 and 12 months
Drug: varenicline
  Arms: varenicline
Drug: placebo
  Arms: placebo

SUMMARY:
Primary aim: Will varenicline be better than placebo to get long-term users of NRT to stop?

Secondary aim: To assess in details some side effects of varenicline i.e. nausea and abnormal dreams.

DETAILED DESCRIPTION:
100-200 long-term users of NRT will be enrolled in a placebo, controlled, randomized trial with varenicline or placebo for 12 weeks to stop the use of NRT.

Assessments consist of carbon monoxide in expired air, p-cotinine, body-weight, questions about craving, nausea and dreams. Primary result is percent not using NRT and not smoking at 12 weeks (point prevalence last 7 days) and secondary result is not smoking and not using NRT at 12 months. Secondary aims, is a more detailed assessment of nausea and dreams; well-known side effects of varenicline and secondary results are a qualitative description of nausea and dreams.

ELIGIBILITY:
Inclusion Criteria:

* Long-term, daily NRT users (except nicotine patch) (>11 months) ex-smokers that are willing to try to stop the use of NRT and adhere to this protocol.
* More than 4 pieces of nicotine gum/ sublingual tablets/ lozenges/ per day, OR more than 3 inhaler cylinders per day, OR
* more than 10 puffs of nasal spray per day.

Exclusion Criteria:

* Age < 18 years,
* CO Smokers,
* Pregnant and lactating women,
* Used varenicline before,
* Not able to cooperate,
* Other significant diseases that might influence the trial (such as moderate -severe cardiac disease, lung cancer,) in expired air > 7 ppm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Primary result is percent not using NRT and not smoking at 12 weeks (point prevalence last 7 days) verified by self-declaration combined with a CO < 8 ppm and a p-cotinine < 15 ng/ml | 12 weeks +/- 1 week

SECONDARY OUTCOMES:
is not smoking and not using NRT at 12 months (point prevalence last 7 days) verified by self-declaration combined with a CO < 8 ppm and a p-cotinine < 15 ng/ml | 12 months +/- 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip Tønnesen, M.D., Principal Investigator — Gentofte Hospital
Locations (1):
- Gentofte Hospital, Copenhagen, Hellerup, Denmark

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Tonnesen P, Mikkelsen K. Varenicline to stop long-term nicotine replacement use: a double-blind, randomized, placebo-controlled trial. Nicotine Tob Res. 2013 Feb;15(2):419-27. doi: 10.1093/ntr/nts146. Epub 2012 Sep 27. PMID 23024246